CLINICAL TRIAL: NCT00703287
Title: Randomized Trial of a Specialized Physiotherapy Program Versus Standard Physiotherapy Advice in Patients With Cervical Dystonia (Spasmodic Torticollis).
Brief Title: Specialized Physiotherapy Program for Cervical Dystonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Donald Grosset (Other)
Collaborators: University of Aberdeen (Other)
Responsible Party: Sponsor-Investigator, Dr Donald Grosset, Consultant Neurologist, South Glasgow University Hospitals NHS Trust
Organization: South Glasgow University Hospitals NHS Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SN07NE039
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-02

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A2 (Sham Comparator): Generic physiotherapy
  Interventions: Other: Physiotherapy
- A1 (Experimental): Specialized Physiotherapy
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Specialized physiotherapy programme developed by Jean-Pierre Bleton
  Other Names: Jean-Pierre Bleton
  Arms: A1
Other: Physiotherapy — Generic physiotherapy
  Arms: A2

SUMMARY:
The investigators wish to establish on a small scale the effectiveness of adding the physiotherapy programme developed by Jean-Pierre Bleton to the present standard treatment for cervical dystonia with a view to undertaking a larger UK-wide trial looking at overall cost-effectiveness. Specifically, the investigators wish to establish:

1. Whether this specific physiotherapy program for cervical dystonia improves patient outcomes in terms of neck position, pain, disability, and quality of life compared to simple physiotherapy advice?
2. What is the minimal clinically important change in the new CDIP-58 quality of life measure for cervical dystonia from a patient's perspective that could then be used to plan a definitive trial of this technique?
3. What are the economic implications of the specialized physiotherapy programme?

ELIGIBILITY:
Inclusion Criteria:

All the following inclusion criteria must be met:

1. Any person over 16 years with primary cervical dystonia causing sufficient interference in lifestyle that they wish to consider physiotherapy treatment and who is able to give informed consent.
2. An abnormal neck position (Toronto Western Spasmodic Torticollis Rating Scale [TWSTR] Part 1A > 0).
3. Patients receiving treatment with botulinum toxin (type A or B) injections (as most will) provided they are on a stable botulinum toxin regimen (i.e. same dose and injection pattern over the previous two injections). This includes those newly diagnosed patients who choose to have botulinum toxin injections OR patients not receiving botulinum toxin (either because of patient preference or previous lack of effect) provided they plan to remain off botulinum toxin for the one year duration of the trial. There will probably be few of these patients but we feel justified in including them because there are no other treatments on offer and because it is presently unknown whether physiotherapy requires botulinum toxin to weaken the muscles in order to have an effect. Anecdotal reports suggest that it can be effective even without botulinum toxin. However, the small numbers who are not receiving botulinum toxin will be analysed as a separate subgroup initially to check whether their response is significantly different to those receiving botulinum toxin.

Exclusion Criteria:

Patients with any of the following criteria will be excluded:

1. Secondary cervical dystonia (e.g. acute onset following trauma or secondary to drugs)
2. A fixed cervical dystonia which may imply a psychogenic component.
3. Radicular or myelopathic features where cervical manipulation may be dangerous.
4. Patients known to have fused cervical vertebrae from previous x-rays
5. Previous use of the Bleton technique.
6. Deep brain stimulation for cervical dystonia.
7. Dementia.
8. Unable to comply with visits for physiotherapy and assessment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To compare different types of physiotherapy for treating condition | Review at 1 month, 3 months & 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Southern General Hospital, 1345 Govan Road, Glasgow, Scotland, United Kingdom